CLINICAL TRIAL: NCT00614146
Title: Therapeutic Impact of Albumin Dialysis With the Molecular Adsorbents Recirculating System (MARS®) in Severely Decompensated Chronic Liver Disease
Brief Title: Recompensation of Exacerbated Liver Insufficiency With Hyperbilirubinemia and/or Encephalopathy and/or Renal Failure
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: 2ConduCT (Industry); G.E.M. mbh Meerbusch (Other); DatInf (Unknown); Gambro Lundia AB (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1438; ISRCTN67377557
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Liver Failure
Keywords: liver failure, albumin dialysis, liver support
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Device: MARS device; Procedure: Standard medical therapy
- 2 (Active Comparator)
  Interventions: Procedure: Standard medical therapy

INTERVENTIONS:
Device: MARS device — 10 treatments with the MARS system during the first three weeks after enrollment of 5-8 hours each.
  Other Names: Liver support
  Arms: 1
Procedure: Standard medical therapy — Standard medical therapy for treatment of the liver disease according to local policy with recommendations as per protocol
  Other Names: SMT
  Arms: 2
Procedure: Standard medical therapy — Standard medical therapy for treatment of the liver disease according to local policy with recommendations as per protocol
  Other Names: SMT
  Arms: 1

SUMMARY:
The objective of this trial is to evaluate the impact of elimination of albumin bound substances during albumin dialysis (MARS®) on mortality and the clinical time course in patients with a recent severe clinical deterioration of chronic liver disease caused by a precipitating (trigger) event within 4 weeks manifested by jaundice, encephalopathy and/or renal failure.

DETAILED DESCRIPTION:
Current medical therapy for end stage liver disease is focused on substitution of blood or plasma products, volume expansion or antibiotic treatment. The only specific treatment is liver transplantation, which is limited by available organs and may be a therapeutic option only for a very minority of patients with recently deteriorated end stage liver disease. The clinical management of defect hepatic synthesis and metabolic regulation has been improved dramatically within the past decades by the development of transfusion and intensive care medicine, but the replacement of detoxification has been more difficult, as the majority of endogenous toxins accumulating in liver failure is bound to albumin. Therefore, conventional dialysis and hemofiltration have been shown to be ineffective for their removal. The present study is based on the theory, that supporting the failing liver by the removal of toxic substances with a biocompatible method (the MARS system) may improve the capacity for recovery of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent by patient or next of kin
* Age greater than 18 years
* Patients with a recent clinical severe decompensation of a presumed cirrhosis (based on clinical evaluation or radiological imaging) related to a precipitating (trigger) event (e.g. infection, bleeding, alcohol abuse)
* Intrahepatic cholestasis (bilirubin greater than 5 mg/dl or greater than 85 µmol/l, respectively) without evidence of extrahepatic origin
* and at least one of the following three:
* Hepatorenal syndrome (impaired renal function with creatinine greater than 1.5 mg/dl or greater than 133µmol/l without evidence of reduced vascular volume [e.g. central venous pressure {CVP} greater than 8 cm H2O] and no evidence of pre-existing renal failure)
* Hepatic Encephalopathy greater than or equal to II°
* Progressive Hyperbilirubinaemia: defined as a more than 50% increase of bilirubin before enrolment, whether in referral or currently in hospital up to a level of greater than 20 mg/dl (or greater than 340 µmol/l)

Exclusion Criteria:

* Progressive jaundice and deterioration as a natural course of a chronic liver disease without precipitating (trigger) event
* Severe thrombocytopenia (platelet count less than or equal to 50 Glutamic Pyruvic Transaminase [GPT]/l)
* Severe coagulopathy (International Normalised Ratio [INR] greater than 2.3)
* Need for renal replacement therapy within three days prior to enrolment
* Severe infection without antibiotic treatment for at least 24 hours. Uncontrolled bacterial infection
* Active bleeding within 48 hours prior to enrolment
* Proven hepatocellular carcinoma (HCC) greater than 4 cm or infiltration of portal vein or acute portal vein thrombosis
* Severe cardiopulmonary disease (New York Heart Association [NYHA] greater than or equal to 2)
* Pregnancy/lactation
* Mean arterial pressure (MAP) less than 60 mmHg despite vasopressor agents (norepinephrine greater than 1 µg/kg/min) for blood pressure support
* Overt clinical evidence for Disseminated Intravascular Coagulation (DIC)
* Clinical evidence for coma of non-hepatic origin
* Extra-hepatic cholestasis
* Severe intrinsic renal disease
* Extended surgical procedure within the last four weeks or unsolved surgical problems
* Known human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2003-04; Primary Completion 2008-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Show improvement of transplant free survival under MARS in comparison to Standard Medical Treatment. | 28 days

SECONDARY OUTCOMES:
Survival regardless of transplantation | 28 days
general survival | 3 months
in-hospital mortality | 3 months
time course of clinical state (number and severity of complications, vital signs, scoring systems, lab tests) | 3 months
economic analysis (length of stay, ICU days, readmissions within observation period) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Banarès, Dr, Study Chair — Hospital Gregorio Maranon, Madrid; Vicente Arroyo, Pf, Study Chair — Clínic Barcelona, Hospital Universitari Villarroel; Roger Williams, Pf, Study Chair — Royal Free and University College Medical School, University College London; Steffen Mitzner, Dr, Study Chair — Dept. of Internal Medicine, University of Rostock
Locations (19):
- AKH Wien, Vienna, Austria
- Universitaire Ziekenhuitzen, Leuven, Belgium
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- France (2):
  - Hôpital Huriez, Lille
  - Hôpital Paul Brousse, Villejuif
- Germany (6):
  - Charite Berlin, Campus Mitte, Berlin
  - Uniklinik Bonn, Bonn
  - Martin Luther Universität Halle-Wittenberg, Halle
  - Klinikum der Universität Regensburg, Regensburg
  - Uniklinik Rostock, Rostock
  - Universitätsklinikum Tübingen, Tübingen
- Catholic University of Rome, Rome, Italy
- Spain (4):
  - Hospital clinic, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital General Universitario, Madrid
  - Hospital Ramon y Cajal, Madrid
- Universitätshospital Zürich, Zurich, Switzerland
- United Kingdom (2):
  - King's College Hospital, London
  - University College London, London

REFERENCES:
- [Background] Stange J, Mitzner S, Ramlow W, Gliesche T, Hickstein H, Schmidt R. A new procedure for the removal of protein bound drugs and toxins. ASAIO J. 1993 Jul-Sep;39(3):M621-5. PMID 8268613
- [Background] Stange J, Ramlow W, Mitzner S, Schmidt R, Klinkmann H. Dialysis against a recycled albumin solution enables the removal of albumin-bound toxins. Artif Organs. 1993 Sep;17(9):809-13. doi: 10.1111/j.1525-1594.1993.tb00635.x. PMID 8240075